CLINICAL TRIAL: NCT01178437
Title: Transcutaneous Non-invasive Stimulation of the Vagus Nerve for the Treatment of Difficult-to-treat Epilepsy - a Prospective Pilot Study Regarding Safety, Effectiveness and Clinical Performance
Brief Title: Transcutaneous Non-invasive Stimulation of the Vagus Nerve for the Treatment of Difficult-to-treat Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: cerbomed GmbH (Industry)
Responsible Party: Chief Medical Officer, cerbomed GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cMPsE01
Record Dates: First submitted 2010-07-29; First posted 2010-08-10 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Epilepsy
Keywords: seizure disorder,; seizures,; convulsions,; grand mal,; petit mal,; absence seizures,; repeated seizures,; children's seizures,; secondary epilepsy,; symptomatic epilepsy,; generalized seizures,; partial seizure,; focal seizure,; partial complex seizure,; anticonvulsant medication
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsy, Tonic-Clonic; Epilepsy, Absence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: T-VNS® Stimulator cM02 (Transcutaneous Stimulation of the Vagus Nerve) — daily, transcutaneous, electrical stimulation of the vagus nerve by the t-VNS device for a period of 9 months
  Other Names: T-VNS® Stimulator cM02

SUMMARY:
The aim of the study is to prove the feasibility and safety of transcutaneous, electrical stimulation of the vagus nerve in patients with difficult-to-treat forms of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Patients of both gender, aged from 18-75 years
* Diagnosis of epilepsy according to the diagnosis criteria of the DSM IV/ ICD 10 (especially G 40.1 /G 40.2/ G 40.3)
* Insufficient response to at least one attempt of treatment in medical history with anticonvulsive medication, dosed sufficiently long and high
* Antiepileptic Drugs (AED) therapy must be stable at a level that promises long-term continuity for at least 10 before study start and has to be continued for at least 3 months during treatment phase

Exclusion Criteria:

* Absence of Informed Consent
* Pregnancy
* Psychiatric diseases, especially post-traumatic stress disorder, obsessive-compulsive disorders, schizophrenia, Borderline personality disorders (BPD), character disorders as well as major depressive disorders, anxiety disorders and eating disorders as comorbidity.
* Abuse of drugs and alcohol until 12 weeks before study start
* Cerebrovascular diseases
* Dementia
* Severe traumatic brain injury in medical history including invasive and non-invasive methods of therapy (tumor surgery, "Gamma Knife Surgery")
* Indications of structural impairment of the basal ganglia or the brain stem
* active implants (e.g. cochlea implants, VNS, pacemaker)
* Severe neurological diseases (e.g. Morbus Parkinson, systemic neurologic diseases
* severe internistic diseases (e.g. arterial hypertension, respiratory failure)
* Bronchial asthma
* malignant diseases of any kind, within five years before study start
* Severe active infectious diseases (e.g. HIV, hepatitis)
* Bone diseases (e.g. Morbus Paget, recent fractures)
* Diseases of the ENT body system: Hearing loss of the left ear which is treated with a hearing instrument, all dermatologic and infectious diseases which affect the area around the pinna and the ear canal, severe malformation of the pinna
* Vagotomy
* Concurrent participation in other studies
* Other circumstances that in the opinion of the investigator might be an obstacle for enrolling the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Assessment of performance | 9 months
  rated by investigator
  QOLIE-89 MADRS CCTE

SECONDARY OUTCOMES:
Patient's subjective assessment of epileptic shocks | 9 months
  rated by patient. Subjective assessment of epileptic shocks and cognitive functions. Measured with "Erlanger Kognitionstest" (EKT)
Further assessment of performance | 9 months
  EEG long-term monitoring, MR spectroscopy
Assessment of Safety | 9 months
  Registration of (S)AEs and drop outs

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Herrmann, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Epilepsiezentrum Erlangen, Erlangen, Bavaria, Germany